CLINICAL TRIAL: NCT02323659
Title: Comparison of Methotrexate Versus Interferon-alfa 2b on Efficacy, Safety and Quality of Life in Patients With Primary Cutaneous T-cell Lymphomas
Brief Title: Comparison of Methotrexate Versus Interferon-alfa 2b in Patients With Primary Cutaneous T-cell Lymphomas
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Polish Lymphoma Research Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PLRG-14
Record Dates: First submitted 2014-12-12; First posted 2014-12-23 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2018-10

CONDITIONS: Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides
Keywords: Mycosis Fungoides; Cutaneous T-Cell Lymphoma; Interferon; Methotrexate
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides | interventions — Methotrexate; Clorazepate Dipotassium; Interferon alpha-2; Introns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methotrexate arm (Active Comparator): Patients assigned to receive methotrexate
  Interventions: Drug: Methotrexate
- Interferon Alfa-2b (Active Comparator): Patients assigned to receive Interferon alfa 2b
  Interventions: Drug: Interferon Alfa-2b

INTERVENTIONS:
Drug: Methotrexate — Methotrexate 20mg per dose, administered orally, once every week
  Other Names: Tranxene
  Arms: Methotrexate arm
Drug: Interferon Alfa-2b — Interferon Alfa-2b 3 million international units (MIU), administered 3 times per week
  Other Names: Intron A
  Arms: Interferon Alfa-2b

SUMMARY:
Comparison of methotrexate versus interferon-alfa 2b on efficacy, safety and quality of life in patients with primary cutaneous T-cell lymphomas after failure of topical or phototherapy treatment.

DETAILED DESCRIPTION:
Methotrexate and interferon are widely used drugs in treatment in patients with cutaneous T-cell Lymphomas. Efficacy and safety of both drugs have never been compared directly in one study.

Patients will be randomly assigned to receive Methotrexate or Interferon Alfa 2b. Treatment will continue until disease progression or the development of intolerable toxicities. Study is conducted to analyse and compare efficacy, safety and quality of life provided by Methotrexate or Interferon Alfa 2b.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed primary cutaneous T-cell lymphoma (CTCL)
2. Age ≥ 18 years
3. Performance status WHO<=2
4. Subject must have adequate bone marrow, renal and hepatic function
5. Topical and phototherapy treatment failure in the past
6. Signed informed consent

Exclusion Criteria:

1. Subject has received prior systemic methotrexate or interferon therapy
2. Unacceptable methotrexate or interferon treatment toxicity in the past
3. Inadequate bone marrow, renal or hepatic function as follows:

   * Bone Marrow: Absolute neutrophil count (ANC) < 1,500/mm 3 (1.5 × 10 9 /L); Platelets <100,000/mm 3 (100 × 10 9 /L); Hemoglobin < 9.0 g/dL (1.4 mmol/L);
   * Renal function: Creatinine >1.5 x Upper limit of normal (ULN)
   * Hepatic function: Aspartate and Alanine transaminase (AST and ALT) >3× ULN; bilirubin > 1.5 × ULN
   * Active hepatitis B or hepatitis C
4. anorexia
5. major depression with suicidal ideation or suicide attempt in the past
6. Symptomatic congestive heart failure
7. Epilepsia or other symptomatic central nervous system dysfunction
8. active skin infection not related to underlying CTCL, active Tuberculosis, HIV infection
9. Subject is pregnant or lactating
10. Psychiatric illness/social situation that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-06-01 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Objective response rate as measured by the modified Severity Weighted Assessment Tool (mSWAT scoring system) | 3 years
  Evaluation according to modified Severity Weighted Assessment Tool (mSWAT scoring system)

SECONDARY OUTCOMES:
Number of Participants With Adverse Events | 3 years
Quality of Life as measured by the Dermatology Life Quality Index (DLQI) | 3 years
  Evaluation according to Dermatology Life Quality Index (DLQI)

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Sokołowska Wojdyło, MD, PhD, Principal Investigator — Polish Lymphoma Research Group; Ewa Chmielowska, MD, PhD, Principal Investigator — Polish Lymphoma Research Group
Locations (1):
- Centrum Onkologii im. prof. F. Łukaszczyka, Bydgoszcz, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956